CLINICAL TRIAL: NCT05240196
Title: Does Actively Listening to Binaural Music Immediately Prior to Mammography Reduce a Patient's Pain Score From Applied Compression During the Procedure
Brief Title: Binaural Music Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tameside General Hospital (Other)
Collaborators: University of Salford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BR/2019/487
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to the following groups;
  1. Control
  2. Binaural music
  3. Non binaural music
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): participant will receive standard care only
- Binaural music (Other): Participants will listen to binaural music whilst having a routine mammogram
  Interventions: Other: music
- Non-binaural music (Other): Participants will listen to non-binaural music whilst having a routine mammogram
  Interventions: Other: music

INTERVENTIONS:
Other: music — playing binaural or non-binaural music
  Arms: Binaural music; Non-binaural music

SUMMARY:
To evaluate client experience relating to mammography and pain scores for patients attending for annual surveillance mammography with a family history of breast cancer. It will involve face to face patient interviews with clients that have had previous mammography at the study site (Tameside and Glossop Integrated Care Trust). The data will be specific to the study site and gathered by the PI only. This is a feasibility study, the data will be used to inform further study across additional sites and application for a College of Radiographers grant. The study is a quantitative assessment of pain following the intervention of binaural music, the mammogram will be undertaken by the same mammographer to standardise technique. Pain will be assessed using a validated numerical 11 point pain score for ease of use as per previous published research.

Each client will feedback twice during the care event:

1. Retrospectively from previous experience
2. Actual pain, if any, during planned mammogram Patients will be randomised to the following groups;

1. Control 2. Binaural music 3. Non binaural music If the feasibility study is successful the study will proceed to a second phase and the number of participants extended to 60 patients per group (180 in total) and the study ceased when the number reached.

If there is an indication to extend to another Trust (multi-site trial). A new IRAS application will be submitted following the feasibility study, if successful.

DETAILED DESCRIPTION:
Principal aim of the study: To investigate whether the experience of mammography-related pain can be improved by listening to binaural music prior to the examination.

The research aims to improve patient experience for patients undergoing annual mammography with moderate or high risk of breast cancer. These patients can commence annual mammography at 40 years of age until entering the National Health Service Breast Screening Program (NHSBSP), (NICE, 2013). Reduction in pain or anxiety for these patients may improve compliance, reduce DNA rates which is a cost saving to the NHS.

Previously, mammography-related pain scores have been evaluated within the study institution in these groups of women by measuring pain using a VAS/NRS pain tool three times; before, immediately after and 1-week post mammography. The results of this study showed that expectation of pain by the patient was the only significant predictor for pain r=0.79. Breast size, compression force, menopausal status and breast density were not found to be significant indicators for pain (Nelson et al., 2018).

One of the action points for this research was to repeat the study within the introduction of a series of pain interventions to improve pain scores for all patients in the low, moderate and severe pain categories.

f. Methodology The feasibility study will be a prospective, randomised controlled trial enabling comparisons based on current pain measurements, for patients attending family history screening at Tameside and Glossop Integrated Care NHS Foundation Trust. If the results are significant then a larger scale study across 2-3 sites is planned.

The patient information sheet (PIS) will be posted with the appointment letter and the patients will have 2 weeks to read the letter and contact the researcher with any questions or concerns prior to their mammogram appointment.

Allocation to the group will be randomised prior to mammogram by selection using an online randomisation tool until the sample size is reached for each group (control, non binaural music, binaural music). The patients will be asked to participate in the study and will not know which group they are in until instructions are given just prior to the examination. The control group will be asked to score their pain before and after routine mammography without actively listening to music.

The patient will be asked to self-evaluate their pain from their most recent previous mammogram from memory using a validated 11-point numerical scale where zero = no pain and 10 = the worst pain. The patient will then be asked to score their pain following their current mammogram and this will be recorded on a second validated 11-point numerical scale (Yale 2018). The information will be recorded by the mammographer for improved consistency and scanned into the radiology information system as a permanent record. The same mammographer will perform the mammograms to standardise technique, the compression given will remain at her discretion. Music will be standardised and played using personal headphones for 5 minutes prior to mammography

ELIGIBILITY:
Inclusion Criteria:

* Bilateral mammogram.
* Asymptomatic patients only.
* Patients attending for family history follow up mammography.
* Patients that have had a mammogram within 2 years at the trust to compare to on the same equipment.
* Patients with language barriers if an interpreter or relative is available.

Exclusion Criteria:

* Patients with mammography elsewhere including screening units or in the private sector.

Family history patients having their 1st mammogram. Patients with breast implants. Patients with inability to consent due to mental incapacity. Patients with hearing impairments Patients with a history of epilepsy Patients with ongoing mental health illness Patients with heart arrhythmia and pacemakers Patients taking prescribed pain medication

Ages: 40 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 57 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Pain score from previous mammography compared with pain score reported at current mammography appointment | pain score collected within 10 minutes post mammograph
  Reported pain score for previous mammography experience compared with the pain score reported for current mammography appointment. Pain will be measured using a validated numerical 11 point pain score scale.

SECONDARY OUTCOMES:
comparison of pain scores reported for each study group | comparison to take place within 3 months post mammography visit
  Correlation statistics will be used to examine trends between prior pain / comfort levels and the new mammography examination following the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Nelson, Principal Investigator — Tameside and Glossop Integrated Care NHS Foundation Trust
Locations (1):
- Tameside and Glossop Integrated Care NHS Foundation Trust, Manchester, United Kingdom